CLINICAL TRIAL: NCT00818389
Title: A Multicenter, Double-Blind, Placebo-Controlled, Study to Investigate the Safety and Efficacy of Lithium in Combination With Riluzole in Volunteers With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Study to Investigate the Safety and Efficacy of Lithium in Volunteers With Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: NINDS DSMB recommended trial be terminated for futility after reviewing an interim analysis of 84 subjects.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ALS Association (Other); ALS Society of Canada (Other Government); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Toronto (Other); State University of New York - Upstate Medical University (Other); Columbia University (Other); University of Kentucky (Other)
Responsible Party: Merit Cudkowicz, MD, MSc, Co-Director, Neurology Clinical Trials Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01NS049640 (NIH); 3U01NS049640-04S1 (NIH)
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; ALS; Lou Gehrig's disease; riluzole; lithium; neurodegeneration
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Nerve Degeneration | interventions — Lithium Carbonate; Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants randomized to lithium/riluzole (randomization is 1:1 lithium/riluzole to placebo/riluzole, i.e., participants have an equal chance of getting randomized to lithium vs. placebo).
  Interventions: Drug: Lithium Carbonate; Drug: Riluzole
- 2 (Placebo Comparator): Participants randomized to placebo/riluzole (randomization is 1:1 lithium/riluzole to placebo/riluzole, i.e., participants have an equal chance of getting randomized to lithium vs. placebo).
  Interventions: Drug: Riluzole; Drug: placebo

INTERVENTIONS:
Drug: Lithium Carbonate — Participants will receive capsules that contain 150 milligrams (mg) lithium carbonate. Participants will be randomized to lithium/riluzole or placebo/riluzole and treated for 52 weeks. Participants originally randomized to placebo who fail (progress) will crossover to lithium for the remainder of the trial.
  Arms: 1
Drug: Riluzole — All participants enrolled in this study will be taking a stable dose of riluzole 50 milligrams (mg) by mouth (PO) twice per day (BID) for at least 30 days prior to screening.
Drug: placebo — an inactive substance
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effectiveness of lithium combined with riluzole to riluzole combined with placebo in people with amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a rare, neurodegenerative disorder that results in progressive wasting and paralysis of voluntary muscles.

In this double blind, randomized, placebo-controlled clinical trial, researchers will evaluate the safety and effectiveness of the drug lithium given in combination with riluzole, a drug commonly used to treat ALS, compared to a placebo given in combination with riluzole.

Approximately 250 participants will be recruited from multiple centers, in the US and Canada, that belong to the Northeast ALS Consortium (NEALS) and the Canadian ALS Clinical Trials and Research Network (CALS). Enrollment will occur in stages. Initially 84 participants will be enrolled in the trial. An interim analysis using available data will occur after the 84th participant is enrolled. During this time, the Data and Safety Monitoring Board (DSMB) appointed by the National Institutes of Health (NIH) may decide to stop the trial for efficacy or futility reasons or to stop enrollment and request that follow-up continue with the 84 participants already enrolled in the trial, or the DSMB may decide to continue enrollment.

Participants will be randomized to one of two arms of the study. Arm one will receive lithium and riluzole. Arm two will receive riluzole and placebo (an inactive substance). All participants will be receiving riluzole. After screening and randomization, participants will be followed every 4 weeks for the first 12 weeks. Subsequent in-person visits will occur every 8 weeks with a final visit at week 52. Between in-person visits, telephone interviews will take place every 4 weeks to administer the Amyotropic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) questionnaire. A follow-up telephone interview will occur at week 56 (off study medication) to review adverse events. The primary outcome measure is disease progression as measured by the ALSFRS-R questionnaire. Participants randomized to placebo whose disease progresses will be crossed over to lithium for the remaining period of the study (up to 52 weeks total).

Duration of the study for participants is 56 weeks which includes 52 weeks of treatment and a followup telephone interview at week 56.

ELIGIBILITY:
Inclusion Criteria:

* Familial or sporadic ALS
* Participants diagnosed with laboratory supported probable, clinically possible, probable or definite ALS according to the World Federation of Neurology Revised El Escorial criteria
* Disease duration from symptom onset no greater than 36 months at the Screening Visit
* Age 18 years or older
* Capable of providing informed consent and complying with trial procedures
* On a stable dose of riluzole 50 milligrams (mg) twice per day(bid) for at least 30 days prior to screening
* Vital capacity (VC) equal to or more than 60% predicted normal value for gender, height and age at the Screening Visit
* Creatinine <1.5 milligrams per deciliter (mg/dl) [133 micromoles per liter (umol/L]
* Participants maintained on thyroid medication must be euthyroid for at least 3 months before the Screening Visit.
* Participants with psoriasis must have inactive disease for at least 30 days before the Screening Visit.
* Women must not be able to become pregnant (e.g., post menopausal for at least one year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. Women of childbearing potential must have a negative serum pregnancy test at the Screening Visit and be non-lactating.
* Geographic accessibility to the study site

Exclusion Criteria:

* History of known sensitivity or intolerability to lithium or to any other related compound
* Prior exposure to lithium within 90 days of the Screening Visit
* Exposure to any investigational agent within 30 days of the Screening Visit
* Participants who are malnourished, dehydrated or on a sodium-free diet will be excluded due to the potential side effects of lithium carbonate
* Use of digoxin or iodide salts [e.g. calcium iodide, hydrogen iodide (hydriodic acid), iodide, iodinated glycerol (Organidin), iodine, potassium iodide (SSKI), and sodium iodide supplementation beyond table salt]
* Presence of any of the following clinical conditions: Substance abuse within the past year; Unstable cardiac, pulmonary, renal, hepatic, endocrine, hematologic, or active malignancy or infectious disease; autoimmune deficiency syndrome (AIDS) or AIDS-related complex; Clinically active psoriasis within 30 days of the Screening Visit; Unstable psychiatric illness defined as psychosis (hallucinations or delusions) or untreated major depression within 90 days of the Screening Visit; Screening serum creatinine greater than or equal to 1.5 mg/dL (133 umol/L), thyroid stimulating hormone (TSH) > 20% above the upper limit; Presence of any clinically significant conduction abnormalities on electrocardiogram (ECG); or Lactating or have a positive serum pregnancy test at the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, MSc, Principal Investigator — Massachusetts General Hospital; Swati Aggarwal, MD, Principal Investigator — Massachusetts General Hospital; Lorne Zinman, MD, MSc, FRCPC, Principal Investigator — Sunnybrook Health Sciences Center, Univ. of Toronto, Toronto, CA; Jinsy Andrews, MD, Principal Investigator — Columbia University, New York, NY
Locations (37):
- United States (22):
  - Phoenix Neurological Assoc., 1331 N. 7th Street, Suite 350, Phoenix, Arizona
  - Cedars-Sinai ALS Center, Neurology Specialty Clinic, 8730 Alden Drive, Thalians, E 245, Los Angeles, California
  - UCSF ALS Center, University of California San Francisco, Neurology, Box 0114, UCSF, San Francisco, California
  - Mayo Clinic-Jacksonville, Neurology Department, 4500 San Pablo Road, Jacksonville, Florida
  - University of Miami, Miller School of Medicine, 1150 NW 14th Street, Suite 609 (SCs are suite 701), Miami, Florida
  - Indiana University, Department of Neurology, 1050 Wishard Blvd, RG 6, Indianapolis, Indiana
  - University of Kentucky Medical Center, BAMC, Department of Neurology, Room A307, 1101 Veteran's Drive, Lexington, Kentucky
  - Johns Hopkins University, Department of Neurology, 600 N. Wolfe St, Meyer 6-181, Baltimore, Maryland
  - Massachusetts General Hospital, 149 13th St, Room 2266, Charlestown, Massachusetts
  - Wayne State University, Department of Neurology, 4201 St. Antoine, 8C UHC, Detroit, Michigan
  - Hennepin County Medical Center, Dept of Neurology, 701 Part Ave S, P5-200, Minneapolis, Minnesota
  - Washington University, 660 S. Euclid Ave., Box 8111 Neurology, St Louis, Missouri
  - Columbia Univ Med Ctr, Eleanor and Lou Gehrig ALS/MDA Center, 710 West 168th St, 9th Floor, New York, New York
  - SUNY Upstate Medical University, 750 E Adams St, 6610UH, Syracuse, New York
  - Duke University Medical Center, Box 3333, Durham, North Carolina
  - Wake Forest University, ALS Center, Paul Sticht Center, Ground Floor, Medical Center Blvd, Winston-Salem, North Carolina
  - Ohio State University, Neuromuscular Division, 1654 Uphan Drive, 417 Means Hall, Columbus, Ohio
  - Penn State Hershey Medical Center, Department of Neurology, H037, Pennsylvania State Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, 245 North 15th Street, Philadelphia, Pennsylvania
  - Texas Neurology, PA, 6301 Gaston Ave, Suite 400 West Tower, Dallas, Texas
  - University of Vermont, Department of Neurology, 89 Beaumont Drive, Given Bldg, Room C-225, Burlington, Vermont
  - University of Virginia, Department of Neurology, 3100 Hospital Drive, Charlottesville, Virginia
- Canada (15):
  - University of Calgary, Area 3, University of Calgary Medical Clinic, 3350 Hospital Drive NW Foothills Hosp. Grounds, Calgary, Alberta
  - University of Alberta, Division of Neurology, Dept of Medicine, 2E3.17 Walter C. MacKenzie Health Sciences Center, Edmonton, Alberta
  - University of British Columbia, GF Strong Rehab Centre, 4255 Laurel Street, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - University of New Brunswick, The Stan Cassidy Centre for Rehabilitation, 800 Priestman St., Fredericton, New Brunswick
  - Dalhousie University, Capital District Health Authority, Queen Elizabeth II Health Sciences Centre, P.O. Box 9000, Summer Street, Halifax, Nova Scotia
  - McMaster University, McMaster University Medical Centre, Hamilton Health Sciences, 1200 Main Street West, Room 4U7, Box 2000, Hamilton, Ontario
  - Queen's University, The Adult Neuromuscular Clinic, PCCC, St. Mary's of the Lake Hospital Site, Department of Physical Medicine and Rehabilitation, 340 Union Street, Postal Bldg 3600, Kingston, Ontario
  - University of Western Ontario, Department of Clinical Neurological Sciences, Motor Neuron Disease Clinic, 339 Windermere Road, Box 5339, London, Ontario
  - University of Ottawa, The Rehabilitation Centre, 505 Smyth Road, Ottawa, Ontario
  - University of Toronto, Sunnybrook Health Sciences Centre, ALS/Neuromuscular Clinic - SCIL, Room UG-35, 2075 Bayview Ave, Toronto, Ontario
  - University of Montreal, CHUM (Centre Hospitalier de l'Université de Montréal) Notre-Dame Hospital 1560,Sherbrooke east street, Montreal, Quebec
  - McGill University, Montreal Neurological Hospital, 3801 University, Room 205, Montreal, Quebec
  - Laval University, CHA-Enfant-Jesus Hospital, 1401, 18th Street, Québec, Quebec
  - University of Saskatchewan, Saskatoon City Hospital, 701 Queen Street, Room 7717 - 7th Floor, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Fornai F, Longone P, Cafaro L, Kastsiuchenka O, Ferrucci M, Manca ML, Lazzeri G, Spalloni A, Bellio N, Lenzi P, Modugno N, Siciliano G, Isidoro C, Murri L, Ruggieri S, Paparelli A. Lithium delays progression of amyotrophic lateral sclerosis. Proc Natl Acad Sci U S A. 2008 Feb 12;105(6):2052-7. doi: 10.1073/pnas.0708022105. Epub 2008 Feb 4. PMID 18250315
- [Derived] Din Abdul Jabbar MA, Guo L, Guo Y, Simmons Z, Pioro EP, Ramasamy S, Yeo CJJ. Describing and characterising variability in ALS disease progression. Amyotroph Lateral Scler Frontotemporal Degener. 2024 Feb;25(1-2):34-45. doi: 10.1080/21678421.2023.2260838. Epub 2024 Jan 23. PMID 37794802
- [Derived] Aggarwal SP, Zinman L, Simpson E, McKinley J, Jackson KE, Pinto H, Kaufman P, Conwit RA, Schoenfeld D, Shefner J, Cudkowicz M; Northeast and Canadian Amyotrophic Lateral Sclerosis consortia. Safety and efficacy of lithium in combination with riluzole for treatment of amyotrophic lateral sclerosis: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2010 May;9(5):481-8. doi: 10.1016/S1474-4422(10)70068-5. Epub 2010 Apr 1. PMID 20363190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2009 to June 2009, 97 patients were screened and 84 subjects were randomized at 21 clinical sites; 11 in the United States and 10 in Canada. All sites were members of the Northeast ALS Consortium (NEALS) and/or the Canadian ALS Consortium (CALS).
Pre-assignment Details: All patients were required to be on a stable dose of riluzole for at least 30 days prior to screening. 13 subjects failed screening: 3 due to low lung function test results, 3 due to prohibited medications,3 due to study closure, 2 due to abnormal lab test results and 1 due to death unrelated to the study.
Groups:
- Lithium + Riluzole: Subjects randomized to lithium + riluzole were required to be taking riluzole 50 milligrams (mg) twice per day at least 30 days prior to the screening visit and during the trial. Lithium carbonate and matching placebo were supplied in 150 mg capsules. Dosing started at 450 mg/day (1 capsule taken in the a.m. and 2 capsules taken in the p.m.), titrated to maintain plasma lithium levels of 0.4 - 0.8 milliequivalent per liter (mEq/L). The number of capsules taken per day was titrated individually for each patient based on blood testing to maintain plasma levels of lithium = 04. - 0.8 milliequivalent per liter (mEq/L).
- Placebo + Riluzole: Participants randomized to placebo + riluzole were required to be taking riluzole 50 milligrams (mg) twice per day at least 30 days prior to the screening visit and during the trial. Matching placebo was supplied in 150 mg capsules. Dosing started at 450 mg/day (1 capsule in the a.m. and 2 capsules in the p.m). Paired sham dosage modifications were made for placebo subjects, i.e. all subjects randomized to placebo were 'paired' with a lithium subject and underwent identical dosage changes to maintain blinding.
Period: Overall Study
Arm/Group | Lithium + Riluzole | Placebo + Riluzole
Started | 40 | 44
Completed | 36 (4 subjects terminated study early before 1st interim analysis. Study terminated early for futility.) | 38 (6 subjects terminated study early before 1st interim analysis. Study terminated early for futility.)
Not Completed | 4 | 6
Not completed — Death | 1 | 3
Not completed — ALS Disease Progression | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium + Riluzole | Placebo + Riluzole | Total
Number analyzed (Participants) | 40 | 44 | 84
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (10.2) | 55.5 (11.9) | 56.24 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 30
  Male | 30 | 24 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 40 | 42 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 39 | 42 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ALS Functional Rating Scale-Revised (ALSFRS-R) [Mean (Standard Deviation); unit: Scores on a scale] — ALSFRS-R is an ordinal rating scale questionnaire (rating 0-4) used to determine subject's assessment of their capability and independence in 12 functional activities (i.e. this is a patient-reported questionnaire scale of disability). Each question has a rating of 0-4 with 4 being the most functional and 0 being the least functional. The most functional total score is 48.
  Scores on a scale | 38.4 (4.6) | 36.5 (5.7) | 37.43 (5.24)
Vital Capacity [Mean (Standard Deviation); unit: Percent of predicted normal] — Vital capacity (VC) testing is a measure of lung function that is performed using a standard spirometer and the Slow VC method. Three trials were required (5 maximum); the best of 3 was used.
  Percent of predicted normal | 94.0 (18.1) | 86.9 (16.9) | 90.18 (18.20)

OUTCOME MEASURES:

1. Secondary Outcome: Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised Questionnaire(ALSFRS-R)
Description: ALSFRS-R is a self-administered ordinal rating scale questionnaire (rating 0-4 for each question,4 is most functional,0-48 total)of 12 functional activities. The most functional total score is 48. ALSFRS-R done at baseline and weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 & 52, dependent on enrollment duration. Secondary efficacy was evaluated by comparing the mean rate of decline of ALSFRS-R score by treatment group.
Time Frame: 9 months: Baseline to study termination (January 2009 - October 2009)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium + Riluzole | Placebo + Riluzole
Number analyzed (Participants) | 40 | 44
Scores on a scale | -1.24 (0.21) | -1.09 (0.20)

2. Primary Outcome: Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised Questionnaire (ALSFRS-R)
Description: ALSFRS-R is a self-administered ordinal rating scale questionnaire (rating 0-4 for each question,4 is most functional,0-48 total)of 12 functional activities. The most functional total score is 48. ALSFRS-R done at baseline and weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 & 52, dependent on enrollment duration. Number of subjects who failed by treatment group was evaluated. Failure was defined as 6-point drop in ALSFRS-R or death from baseline.
Time Frame: 9 months: Baseline to study termination (January 2009 - October 2009)
Measure: Number; unit: Participants
Arm/Group | Lithium + Riluzole | Placebo + Riluzole
Number analyzed (Participants) | 40 | 44
Participants | 18 | 14

3. Secondary Outcome: Vital Capacity (VC) (Percent of Predicted Normal)
Description: Secondary efficacy was measured by comparing the rate of decline of mean VC by treatment group.
Time Frame: 9 months: Baseline to study termination (January 2009- October 2009)
Measure: Mean (Standard Error); unit: Percent of predicted normal
Arm/Group | Lithium + Riluzole | Placebo + Riluzole
Number analyzed (Participants) | 40 | 44
Percent of predicted normal | -1.89 (0.45) | -3.12 (0.47)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study period: January 2009 to October 2009. Each subject was followed for AEs from consent signing to the end of their study participation. The AEs reported here are treatment emergent AEs.
Description: The study was terminated early after the first interim analysis for futility. The first interim analysis was conducted in September 2009. The first subject was randomized in January 2009 and the last follow-up for study subjects was in October 2009.
Arm/Group | Lithium + Riluzole | Placebo + Riluzole
Serious Adverse Events (participants affected / at risk) | 10/40 | 8/44
Other Adverse Events (participants affected / at risk) | 39/40 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium + Riluzole (N=40) | Placebo + Riluzole (N=44)
Benign tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) — Secondary to suspected pulmonary embolism
Cardiac pain (Cardiac disorders) | 0 (0) | 1 (1)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chest/thorax pain (General disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) — Depression with suicide attempt
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Nervous system disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hemorrhage, CNS (Nervous system disorders) | 1 (1) | 0 (0) — Traumatic subdural hematoma
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Retro-orbital pain (Eye disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Speech impairment/dysphagia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope/fainting (Nervous system disorders) | 1 (1) | 0 (0)
Thrombosis/embolism (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium + Riluzole (N=40) | Placebo + Riluzole (N=44)
Anorexia (Gastrointestinal disorders) | 6 (7) | 2 (4)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Blood and lymphatic system disorders) | 5 (7) | 1 (2)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (7) | 8 (9)
Depression (Psychiatric disorders) | 6 (9) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 5 (6)
Dizziness (Nervous system disorders) | 5 (6) | 1 (1)
Drooling (Gastrointestinal disorders) | 7 (7) | 6 (7)
Dysarthria/voice changes (Nervous system disorders) | 7 (7) | 4 (5)
Dysphagia (difficulty swallowing) (Nervous system disorders) | 6 (9) | 9 (9)
Dysphasia/speech impairment (Nervous system disorders) | 4 (5) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 6 (10)
Edema (limb) (Blood and lymphatic system disorders) | 6 (12) | 7 (8)
Fall (Nervous system disorders) | 8 (17) | 2 (7)
Fasciculations (Nervous system disorders) | 7 (12) | 4 (7)
Fatigue (General disorders) | 14 (24) | 9 (13)
Headache (General disorders) | 7 (7) | 8 (11)
Heartburn (Gastrointestinal disorders) | 4 (5) | 5 (6)
Infection (sinus) (Infections and infestations) | 3 (5) | 1 (1)
Infection (upper airway) (Infections and infestations) | 4 (6) | 3 (3)
Insomnia (Nervous system disorders) | 5 (5) | 5 (5)
Joint pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 7 (8)
Muscle atrophy (wasting) (Nervous system disorders) | 3 (3) | 2 (7)
Muscle cramps (Nervous system disorders) | 4 (5) | 3 (4)
Muscle weakness (facial) (Nervous system disorders) | 2 (2) | 2 (3)
Muscle weakness (generalized) (General disorders) | 4 (8) | 7 (10)
Muscle weakness (lower extremity) (Nervous system disorders) | 16 (25) | 17 (29)
Muscle weakness (trunk) (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4)
Muscle weakness (upper extremity) (Nervous system disorders) | 20 (24) | 17 (25)
Nausea (Gastrointestinal disorders) | 10 (14) | 9 (13)
Pain (back) (Musculoskeletal and connective tissue disorders) | 6 (10) | 1 (1)
Pain (chest) (General disorders) | 4 (5) | 2 (2)
Pain (extremity) (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (6) | 0 (0)
Pyramidal tract dysfunction (increased muscle tone and/or brisk reflexes) (Nervous system disorders) | 8 (9) | 3 (4)
Somnolence (Nervous system disorders) | 2 (2) | 2 (3)
Stomach discomfort (Gastrointestinal disorders) | 2 (5) | 0 (0)
Tremor (Nervous system disorders) | 6 (7) | 3 (3)
Urinary frequency/urgency (Renal and urinary disorders) | 7 (9) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (5)
Weight loss (General disorders) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No